CLINICAL TRIAL: NCT06611124
Title: Surgical Evaluation of Fixation of Hand Metacarpals Fractures With K-wires
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Ali Helmi (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ali Helmi, aasitant professor in faculty of medicine ,sohag universty, Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-05-01MD
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Metacarpal Fracture

STUDY DESIGN:
Intervention Model Description: reduction with axial traction to disimpact the fracture with dorsal pressure for metacarpals shfat and head fractures pinng of the fracture with k-wire for fixation
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- k -wires (Other): fixation of hand metacarpals fractures with k-wire 2 arms
  Interventions: Procedure: k -wires fixation for metacarpals fractures
- k -wire (Other): fixation of hand metacarpals fractures with k-wire 2 arms
  Interventions: Procedure: k -wires fixation for metacarpals fractures

INTERVENTIONS:
Procedure: k -wires fixation for metacarpals fractures — reduction and fixation of metacarpal fracture with k-wire

SUMMARY:
different techniques have been described forfracture fixation ofmetacarpals fracture withk-wires being the most described technique as it is minimally invasive methodsfor metacarpals fractures in this research ,we are aimingto evaluate k-wire fixation of metacarpal fracture to optimize the clical outcome as regardsto the degree of stiffnessas avouding the impairment of the gluding tissue of the fingers

DETAILED DESCRIPTION:
hand fractures is about 19%of all fractures k-wires fixation is the most frequently method operative procedure which provide operative stability,early mobilization and excellent functional results primary option for fixation of theses fractures include k-wires ,plateand screws and more recently headless intramedullay compression scres and Bouquet k -wire technique Aim of work fir evaluation of the clinical,functional and radiological outcome of metacarpals fractures fixed by k -wires with variious techniques as antigrade intramedullay k-wires,transverse pinning of unstable displaced shaft and neck fractures.

also direct orif for intra articular head fractures Materials and Methods we are analyzing all patients with metacarpals fractures except patients abnormal hands fuctions before injury procedure done under general anesthesia ,brachial plexus block and wrist block outcome and evaluation handgrip strength 3 month after surgery Geniometer for range of motion AP ,Lateral and oblique radiograph

ELIGIBILITY:
Inclusion Criteria:

* all patients with metacarpal fracture

Exclusion Criteria:

* patients with abnormal hand function before surgery

Min Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
hand grip by goniometer | one year
  hand grip by goniometer

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mohamed Ali Helmi Farghali, Sohag, Asyut Governorate
  - Mohamed Ali Helmi, Sohag

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geissler WB. Operative fixation of metacarpal and phalangeal fractures in athletes. Hand Clin. 2009 Aug;25(3):409-21. doi: 10.1016/j.hcl.2009.05.005. PMID 19643340
- [Result] Kozin SH, Thoder JJ, Lieberman G. Operative treatment of metacarpal and phalangeal shaft fractures. J Am Acad Orthop Surg. 2000 Mar-Apr;8(2):111-21. doi: 10.5435/00124635-200003000-00005. PMID 10799096
- [Result] Moore A, Varacallo MA. Metacarpal Hand Fracture (Archived). 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536960/ PMID 30725645